CLINICAL TRIAL: NCT06408623
Title: A Phase II Clinical Study on the First-line Treatment of Advanced Liver Cancer With Chidamide Combined With Sintilimab and Bevacizumab
Brief Title: Chidamide Combined With Sintilimab and Bevacizumab for the First-line Treatment of Advanced Liver Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q75
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: chidamide combined with Sintilimab and bevacizumab

INTERVENTIONS:
Drug: chidamide combined with Sintilimab and bevacizumab — chidamide combined with Sintilimab and bevacizumab

SUMMARY:
The purpose of this study is to explore the safety and tolerability of chidamide in combination with Sintilimab and bevacizumab in patients with advanced liver cancer, to determine the recommended dose for this combination regimen, and to explore preliminary efficacy data. And based on the tumor immune microenvironment multidimensional (lymphocyte subsets, multiple cytokines, multicolor fluorescence immunohistochemistry, single cell sequencing, etc.) to explore the therapeutic efficacy related markers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old and ≤75 years old, regardless of gender;
* 2. Hepatocellular carcinoma confirmed by histology or cytology;
* 3. Have not received any previous systematic therapy for HCC;
* 4. Barcelona (BCLC) has stage B-C and is not suitable for surgical local treatment, or progresses after surgery and/or local treatment;
* 5. Child-Pugh liver function grade A and good grade B (≤7 points)
* 6. ECOG score 0-1;
* 7. Have at least one measurable lesion (according to RECIST v1.1 assessment criteria);
* 8. Expected survival time ≥3 months;
* 9. The functional level of vital organs must meet the requirements before the first use of the experimental drug; (1) Blood system function (no blood transfusion and no cell growth factor correction within 14 days before screening) : neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109/L, hemoglobin ≥ 90 g/L; (2) Liver and kidney function (no albumin infusion within 14 days before screening) : serum total bilirubin ≤ 1.5 times the upper limit of normal (ULN), serum albumin ≥ 29 g/L, ALT and AST ≤ 2.5×ULN; Serum creatinine ≤1.5×ULN or endogenous creatinine clearance (Cockcroft-Gault formula) ≥60ml/min; (3) Coagulation function: International standardized ratio (INR) ≤1.5 or prothrombin time (PT) exceeding the normal control range ≤6 seconds; (4) Left ventricular ejection fraction (LVEF) ≥ 50% by two-dimensional echocardiography;
* 10. Subjects (both female and male) agree to use effective contraceptive methods for contraception from the date of signing the informed consent to 180 days after the last use of the experimental drug. A woman of childbearing age cannot be pregnant or lactating;
* 11. Patients with active hepatitis B infection who had HBV DNA<2000 IU/ml during the 28 days prior to study entry and who were receiving treatment and taking stable doses of antiviral drugs for at least 7 days upon study entry;
* 12. Any acute, clinically significant treaty-related toxicity must be restored to ≤ grade 1 (according to CTCAE v5.0) prior to initial use of the investigational drug, except for hair loss;
* 13. Voluntarily participate in this clinical trial and sign a written informed consent.

Exclusion Criteria:

* 1. Imaging examination showed that large intrahepatic hemangioma thrombus was complicated (including synchronous thrombus of main portal vein and left and right branches, synchronous thrombus of main portal vein and superior mesenteric vein, and inferior vena cava thrombus);
* 2. Subjects with symptomatic central nervous system (CNS) metastases are not admitted. Subjects with a history of treated CNS metastases (surgical treatment or radiotherapy) were not eligible for inclusion unless they were stable for ≥4 weeks after treatment and had stopped systemic sex hormone therapy (at any dose) for > 2 weeks;
* 3. Patients who had clinically uncontrollable pleural effusion, peritoneal effusion, pericardial effusion, etc. before receiving the study for the first time and could not be enrolled by the researchers. ;
* 4. Patients with a history of other malignancies within 5 years prior to signing informed consent (except cured basal cell skin cancer, skin squamous cell carcinoma, and/or carcinoma in situ after radical resection)
* 5. Active autoimmune disease that may worsen in the course of receiving investigational drug therapy
* 6. In the judgment of the investigator, there are conconitant diseases that seriously threaten the safety of the subjects or affect the completion of the study, such as hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg) that cannot be controlled by two or more antihypertensive drugs, and diabetes that is not well controlled;
* 7. History of hypertensive crisis or hypertensive encephalopathy
* 8. The presence of disease requiring systemic treatment with corticosteroids (>10 mg daily or equivalent of prednisone) or other immunosuppressive agents within 2 weeks prior to initial study treatment
* 9. History of allogeneic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation)
* 10. Systemic infections or other serious infections requiring intravenous antibiotic treatment >7 days within 2 weeks prior to first use of the experimental drug
* 11. HIV positive; HCV antibody positive and HCV RNA positive [Note: if the HCV RNA test result is negative, it can be considered not infected with HCV]; Patients with co-infection of HBV and HCV
* 12. People who are known to have received anti-tuberculosis therapy within one year prior to first receiving study therapy
* 13. Subjects with any of the following cardiovascular diseases were excluded: a) acute myocardial infarction occurred within 6 months prior to first administration of the investigational drug. b) Past and/or current New York Heart Association Class III or IV heart failure. c) Currently has poorly controlled cardiovascular disease, including angina, pulmonary hypertension, or severe heart rhythm or conduction abnormalities. d) Prior to first administration of the trial drug, the 12-lead ECG showed an average QT interval (QTcF) of >450 ms (male) or >470 ms (female).
* 14. The patient is known to have a history of psychotropic substance abuse, alcohol abuse or drug use; A clear history of neurological or psychiatric disorders, including epilepsy or dementia or hepatic encephalopathy.
* 15. People who have participated in other clinical studies and used other clinical trial drugs within 4 weeks before using the experimental drug.
* 16. Previously received immunotherapy, including immune checkpoint inhibitory antibodies (such as anti-PD-1, PD-L1, CTLA-4 antibodies, etc.), immune checkpoint activating antibodies (such as: Anti-icos, CD40, CD137, GITR, OX40 antibody, etc.), and immune cell therapy, or have previously received anti-VEGF, VEGFR targeted therapy or HDACi therapy.
* 17. Chinese patent medicine treatment: Subjects who had received Chinese patent medicine for primary liver cancer before enrollment could be enrolled only after 4 weeks of elution, and the use was prohibited during the trial.
* 18. The patient is known to have a prior allergy to macromolecular protein preparations, or to any investigational drug component.
* 19. Live vaccine was administered within 4 weeks prior to the first administration of the experimental drug.
* 20. Underwent major surgery within 4 weeks prior to the first use of the investigational drug or anticipated major surgery during the study period.
* 21. Persons with past or current interstitial lung disease, coniosis, radiation pneumonia, severe impairment of lung function, etc. that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
* 22. Patients with a history of hemoptysis (i.e., coughing up at least 1/2 TSP (2.5ml) of bright red blood) or a history of gastrointestinal bleeding within 2 months prior to the first use of the trial drug who were judged by the investigator to be ineligible for admission.
* 23. Presence of intestinal obstruction and/or previous clinical signs or symptoms of gastrointestinal obstruction prior to initial use of the investigational drug. Subjects with symptoms and signs of incomplete obstruction/obstruction at initial diagnosis who are treated and whose symptoms have resolved may be enrolled upon investigator assessment.
* 24. Major vascular disease (e.g., aortic aneurysms requiring surgical repair or recent peripheral arterial thrombosis) occurred 6 months before the first use of the investigational drug.
* 25. Evidence of bleeding tendency and major clotting disorder.
* 26. Previous history of intracranial or spinal bleeding; Patients with a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding or portal hypertension within 6 months prior to the first use of the investigatory drug, and patients considered to be at high risk of bleeding (including moderate to severe esophageal and gastric varices at risk of bleeding, locally active gastrointestinal ulcers, and persistent positive fecal occulting blood), should undergo gastroscopy. Patients with "red sign" were excluded.
* 27. Severe open wounds or active peptic ulcers or untreated fractures prior to first use of the experimental drug.
* 28. Current or recent (within 10 days prior to first administration) treatment with aspirin (> 325 mg/ day), clopidogrel (> 75mg/ day) or current or recent treatment with dipyridamole, ticlopidine, and ciliostazole; Therapeutic anticoagulant therapy (except low molecular weight heparin) was used within 2 weeks prior to enrollment.
* 29. Patients who, in the judgment of the investigator, may increase risks associated with the study, may interfere with the interpretation of the study results, or who are deemed unsuitable for enrollment by the investigator and/or sponsor.
* 30. Abdominal or bronchoesophageal fistula, gastrointestinal perforation, or internal abdominal abscess developed within 6 months prior to first administration of the experimental drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months
  progression free surival